CLINICAL TRIAL: NCT01860092
Title: New Enrollment Post-Approval Study of the Argus® II Retinal Prosthesis System
Status: Terminated | Type: Observational
Why Stopped: Manufacturing ceased for all Argus II and Argus 2s devices (FDA notified of and subsequently approved discontinuation of post approval study in Oct 2021)
Sponsor: Second Sight Medical Products (Industry)
Responsible Party: Sponsor
Other Study IDs: PM-02
Record Dates: First submitted 2013-05-14; First posted 2013-05-22 (Estimated); Last update posted 2021-12-23 (Actual); Status verified 2021-12

CONDITIONS: Retinitis Pigmentosa
MeSH Terms: conditions — Retinitis Pigmentosa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | US Export: No

GROUPS / COHORTS (1):
- Argus II Retinal Prosthesis: Patients implanted with the Argus II Retinal Prosthesis

SUMMARY:
This post-approval study is being implemented to monitor the use of Argus II System in a larger US population than available within pre-approval studies. An attempt will be made to include all eligible and willing subjects implanted with Argus II System in the United States.

DETAILED DESCRIPTION:
Safety data will be monitored to ensure continued acceptability of risks to study subjects. The utility (i.e. visual function and functional vision) and reliability of Argus II System will also be evaluated.

There is no study hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* Are adults, age 25 year or older;
* Have severe to profound retinitis pigmentosa;
* Bare light or no light perception in both eyes; if the patient has no residual light perception, then evidence of intact inner layer retina function must be confirmed;
* Have previous history of useful form vision.
* Aphakic or pseudophakic. (If the patient is phakic prior to implant, the natural lens will be removed during the implant procedure.)
* Patients who are willing and able to receive the recommended post-implant clinical follow-up, device fitting, and visual rehabilitation;
* Have consented to the implantation of an Argus II Retinal Prosthesis and subsequently consent to participate in this study;
* At the time of the Baseline Visit, do not suffer from non-ophthalmic serious adverse events (e.g. myocardial infarction, etc.) and

Exclusion Criteria:

* Ocular diseases or conditions that could prevent Argus II System from working (e.g. optic nerve disease, central retinal artery or vein occlusion, history of retinal detachment, trauma, severe strabismus);
* Ocular structures or conditions that could prevent the successful implantation of the Argus II Implant or adequate healing from surgery (e.g. extremely thin conjunctiva, axial length <20.5 mm or >26 mm, corneal ulcers, etc.);
* Ocular diseases or conditions (other than cataracts) that prevent adequate visualization of the inner structures of the eye (e.g. corneal opacity, etc.);
* Inability to tolerate general anesthesia or the recommended antibiotic and steroid regimen associated with the implantation surgery;
* Metallic or active implantable device(s) (e.g. cochlear implant) in the head;
* Pre-disposition to eye rubbing;
* Any disease or condition that prevents understanding or communication of informed consent, study demands, and testing protocols, including:

  * cognitive decline including diagnosed forms of dementia and/or progressive neurologic disease,
  * psychiatric disease including diagnosed forms of depression;
  * does not speak a principal language associated with the region, and
  * deafness;
* Pregnant or wish to become pregnant during the course of the study;
* Participating in another investigational drug or device study that may conflict with the objectives, follow-up or testing of this study;
* Conditions likely to limit life to less than 1 year from the time of inclusion.

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Age 25 years or older; both males and females; with severe to profound retinitis pigmentosa; with bare or no light perception in both eyes or with retinal response to electrical stimulation; with previous history of useful form vision
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2014-01; Primary Completion 2020-03 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
Safety subjects have reached 2 years post-implant. | 5 Years
  Adverse event rates with the main safety analysis performed when all visits completed

SECONDARY OUTCOMES:
Visual function | 5 Years
  Visual function means how to the eye works (e.g. visual acuity). Visual function will be measured using the following test: Square Localization, Direction of Motion and Grating Visual Acuity (GVA).In addition to these tests, a photographic flash test will be performed with the System OFF only to determine if subjects' native residual vision is bare light perception or no light perception.
Functional Vision | 5 Years
  Functional vision means how subjects perform in vision-related activities of daily living. Function vision will be assessed using the Functional Low-Vision Observer Rated Assessment (FLORA). A utilization questionnaire will also be administered to track how subjects are using the Argus II System.
Device Reliability | 5 Years
  Device reliability will be measured by calculating the rate of implant failure over time.

CONTACTS AND LOCATIONS:
Overall Officials: Jessy Dorn, PhD, Study Director — Second Sight Medical Products, Inc.
Locations (17):
- United States (17):
  - University of Southern California, Los Angeles, California
  - University of Colorado, Denver, Denver, Colorado
  - U. of Miami, Bascom Palmer Eye Institute, Miami, Florida
  - University of Miami Bascom Palmer Eye Institute, Miami, Florida
  - Emory University, Atlanta, Georgia
  - Retina Consultants of Hawaii, ‘Aiea, Hawaii
  - University of Illinois at Chicago, Chicago, Illinois
  - Johns Hopkins, Lions Vision Center, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - University of Michigan, Kellogg Eye Center, Ann Arbor, Michigan
  - University of Minnesota Department of Ophthalmology, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Stony Brook University, East Setauket, New York
  - Duke University Eye Center, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Wills Eye Hospital / Mid Atlantic Retina, Philadelphia, Pennsylvania
  - Retina Foundation of the Southwest, Dallas, Texas

REFERENCES:
- [Derived] Yue L, Wuyyuru V, Gonzalez-Calle A, Dorn JD, Humayun MS. Retina-electrode interface properties and vision restoration by two generations of retinal prostheses in one patient-one in each eye. J Neural Eng. 2020 Apr 9;17(2):026020. doi: 10.1088/1741-2552/ab7c8f. PMID 32131056
- [Derived] Gregori NZ, Callaway NF, Hoeppner C, Yuan A, Rachitskaya A, Feuer W, Ameri H, Arevalo JF, Augustin AJ, Birch DG, Dagnelie G, Grisanti S, Davis JL, Hahn P, Handa JT, Ho AC, Huang SS, Humayun MS, Iezzi R Jr, Jayasundera KT, Kokame GT, Lam BL, Lim JI, Mandava N, Montezuma SR, Olmos de Koo L, Szurman P, Vajzovic L, Wiedemann P, Weiland J, Yan J, Zacks DN. Retinal Anatomy and Electrode Array Position in Retinitis Pigmentosa Patients After Argus II Implantation: An International Study. Am J Ophthalmol. 2018 Sep;193:87-99. doi: 10.1016/j.ajo.2018.06.012. Epub 2018 Jun 27. PMID 29940167